CLINICAL TRIAL: NCT00952107
Title: Objective Flap Assessment During Reconstructive Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, John V. Frangioni, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2009P-000095/1; BIDMC
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Cancer
Keywords: breast cancer; breast reconstructive surgery; flap assessment
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging system operation (Experimental)
  Interventions: Device: FLARE imaging system

INTERVENTIONS:
Device: FLARE imaging system — Testing of operation of imaging system

SUMMARY:
The main purpose of this study is to test the ergonomics of an investigational imaging system that can take pictures of blood vessels under the skin. In plastic and reconstructive surgery, blood flow to tissue determines whether the tissue can be transplanted from one location to another. This new imaging device uses invisible near-infrared fluorescent light to see blood vessels that otherwise could not be seen by eye. This study will test the system's basic operation and ergonomics in the operating room.

DETAILED DESCRIPTION:
To perform a pilot study of the FLARE™ NIR fluorescence imaging system in conjunction with indocyanine green (ICG) during breast reconstructive surgery utilizing deep inferior epigastric perforator (DIEP) flaps.

Due to patient-to-patient anatomic variation, the vascular perfusion to the cutaneous elements in flaps is unpredictable and of great concern to the surgeon planning the design of the flap. We propose a method of imaging the flap based on the use of invisible near-infrared fluorescent light that has significant advantages for both patient and surgeon.

Specific Aims:

A pilot optimization study of the imaging system in combination with ICG to determine optimal dose, light excitation fluence rate, and camera exposure time.

ELIGIBILITY:
Inclusion Criteria:

* Women or men above the age of 21 who are undergoing unilateral breast reconstruction after mastectomy.
* Women of childbearing age must have a negative pregnancy test as confirmed by anesthesiologist.

Exclusion Criteria:

* Patients with a known or suspected iodide or seafood allergy.
* Patients with known renal, cardiac, hepatic, or pulmonary disease.
* BMI > 30

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
System operation | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: John V Frangioni, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lee BT, Hutteman M, Gioux S, Stockdale A, Lin SJ, Ngo LH, Frangioni JV. The FLARE intraoperative near-infrared fluorescence imaging system: a first-in-human clinical trial in perforator flap breast reconstruction. Plast Reconstr Surg. 2010 Nov;126(5):1472-1481. doi: 10.1097/PRS.0b013e3181f059c7. PMID 21042103
- See also: Principal Investigator's website — http://www.frangionilab.org